CLINICAL TRIAL: NCT02591446
Title: Transcranial Magnetic Stimulation Studies in Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: Nancy Lurie Marks Family Foundation (Other); Bradley Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 413114
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability
Keywords: TMS; Autism Spectrum Disorders; Plasticity
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Autism Spectrum Disorder (ASD) is the most prevalent of the developmental disorders and their incidence is rising. However, the variability in the behavioral symptoms is large. In part for these reasons, the ASD clinical diagnosis is challenging and often is not made until 3-5 years of age. Thus, there remains an unmet need for a valid and reliable marker which would facilitate ASD diagnosis early in life, enable efficient study of ASD risk factors, and eventually serve as a useful marker to inform the development of effective therapies and assess treatment response in future clinical trials. The specific brain based marker that investigators are currently evaluating is brain plasticity (the changes that occur in your brain through experience). Investigators measure brain plasticity using noninvasive brain stimulation including transcranial magnetic stimulation (TMS) combined with brain imaging, EEG, and behavioral outcome measures. Their work to date demonstrates the potential utility of these techniques in higher-functioning adolescents and adults with ASD, and pilot data support the feasibility and safety of applying the same measures to children and lower functioning individuals.

In this study, investigators will evaluate the validity of this marker in low- and high-functioning adults with ASD, in low- and high-functioning children with ASD, and assess the reliability of this marker.

DETAILED DESCRIPTION:
The clinical, social and financial burden of Autism Spectrum Disorder (ASD) is staggering. They are the most prevalent of the developmental disorders and their incidence is rising. However, the ASD phenotype variability is large, and ASD symptoms can manifest over a range of ages and to different degrees. In part for these reasons, the ASD clinical diagnosis is challenging and often is not made until 3-5 years of age. Thus, there remains an unmet need for a valid and reliable endophenotype which would facilitate ASD diagnosis early in life, enable efficient study of ASD risk factors, and eventually serve as a useful biomarker to inform the development of effective therapies and assess treatment response in future clinical trials. The overarching goal of this proposal is to explore the utility of transcranial magnetic stimulation (TMS) measures of brain plasticity as a novel neurophysiologic endophenotype in high- and low-functioning adults and children with ASD.

Investigators' work to date demonstrates the potential utility of these measures in higher-functioning adults with ASD, and pilot data support the feasibility and safety of applying the same measures to children and lower functioning individuals in whom the value of such an endophenotype would be particularly high. Investigators thus propose to apply single-pulse TMS to evaluate the modulation in corticospinal reactivity induced by a specific repetitive TMS protocol known as theta burst stimulation (TBS). The comparison of the motor responses induced by single-pulse TMS before and following TBS is a unique noninvasive measure of brain plasticity in humans, and investigators have found that it shows a reliable abnormality in high-functioning adult individuals with ASD.

Each subject's participation in the study will consist of three visits: a screening visit and two identical study visits 1-3 weeks apart. Each visit will last for approximately 2 hours. During the first study visit the participants will provide informed consent. patients will then receive a thorough medical history and neurological and physical exam by a licensed physician with training in pediatric medicine. This will evaluate for underlying neurological disorders that would be exclusionary (e.g. motor impairments, epilepsy, medication contraindications etc.) All subjects will also complete a neuropsychological evaluation including IQ and ASD specific evaluations. If eligible to continue, the participant will then return within two weeks to undergo the first TMS evaluation. The TMS procedure will then be repeated 1-3 weeks later. The two identical TMS study visits aim to address reliability of the TMS-based measures: Investigators hypothesize that the TMS measures will be consistent across sessions within all study groups (ASD and controls, adults and children, low- and high-functioning individuals). Such test-retest reliability data are critical to explore the utility of the TMS measures as a potential marker for diagnosis and therapeutic efficacy of an intervention. Investigators thus anticipate that data from the proposed studies will address an important need for a rapid, noninvasive, reliable and safe endophenotype available to patients with ASD across ages and level of function.

ELIGIBILITY:
Inclusion Criteria:

* For ASD group: Clinical diagnosis of a disorder on the autism spectrum according to:

  1. DSM 5 criteria
  2. Assessment using the Autism Diagnostic Interview-Revised
  3. Autism Diagnostic Observation Schedule.
* For the Control group:

  1. No history of ASD or other developmental delay
  2. No history of ASD or other developmental delay in first degree relatives.
* For the group of individuals with Intellectual Disability: Mild to moderate intellectual disability with IQ < 70, but with no ASD.
* Age range: 6-45
* IQ: High functioning individuals will have an IQ>90; Low functioning individuals will have an IQ < 70 with mild-moderate intellectual disability.
* Informed consent (and if needed parental assent).

Exclusion Criteria:

* Intracranial pathology, cerebral palsy, history of severe head injury, or significant dysmorphology;
* History of fainting spells of unknown or undetermined etiology that might constitute seizures;
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy;
* Any progressive (e.g., neurodegenerative) neurological disorder;
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.);
* Metal implants (excluding dental fillings);
* Pacemaker;
* Implanted medication pump;
* Vagal nerve stimulator;
* Deep brain stimulator;
* TENS unit (unless removed completely for the study);
* Ventriculo-peritoneal shunt;
* Signs of increased intracranial pressure;
* Intracranial lesion (including incidental finding on MRI);
* History of head injury resulting in prolonged loss of consciousness;
* Substance abuse or dependence within the past six months;
* Chronic treatment with prescription medications that decrease cortical seizure threshold
* Pregnancy
* Control participants will be excluded from taking part in the study if they have diagnosis of psychiatric condition and if they have family history for ASD.

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will study a total of 120 individuals with ASD. We will also evaluate a total of 120 controls. Ages 6 - 45
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Motor Evoked Potential | Immediately following TMS Motor Threshold determination.
  Motor Evoked Potential will be assessed using electromyogram (EMG). The computer data will be de-identified.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Oberman, PhD, Principal Investigator — Lifespan
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States